CLINICAL TRIAL: NCT04624217
Title: A Phase Ib/II Trial of SHR-1701 Combined With Gemcitabine and Albumin Paclitaxel in First-line Treatment of Subjects With Advanced/Metastatic Pancreatic Cancer
Brief Title: A Trial of SHR-1701 in Combination With Gemcitabine and Albumin Paclitaxel in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-II-204
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — SHR-1701; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1701 (Experimental): SHR-1701 in Combination With Gemcitabine and Albumin Paclitaxel
  Interventions: Drug: SHR-1701

INTERVENTIONS:
Drug: SHR-1701 — PDL1/TGFβ
  Other Names: Gemcitabine and Albumin Paclitaxel

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and tolerability of SHR-1701 in combination with gemcitabine and albumin paclitaxel in first-line treatment of subjects with advanced/metastatic pancreatic cancer, and determine the RP2D for SHR-1701 in the combined regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 70 years;
* Life expectancy ≥ 12 weeks judged by the investigator.
* The ECOG performance status was 0-1.
* At least 1 measurable lesion conforming to RECIST 1.1 criteria.
* In subjects with histologically or cytologically confirmed pancreatic cancer, there was evidence of inoperable locally advanced or distant metastases.
* Adequate organ and bone marrow function.
* Female subjects of childbearing age must undergo a serum pregnancy test within 7 days before the commencement of the study and the results are negative, and are willing to use a medically approved high potency contraceptive method during the study period and within 3 months after the last administration of the study drug; For male subjects whose partner is a female of childbearing age, they should be surgically sterilized or agree to use an effective method of contraception during the study period and for 3 months after administration of the last study.
* Willing to consent and signed the informed consent, and able comply with the planned visit, research treatment, laboratory examination and other test procedures.

Exclusion Criteria:

* Known allergy to the study drug or any of its excipients; Or had a serious allergic reaction to other monoclonal antibodies.
* Previous exposure to drugs/antibodies acting on T cell co-stimulation or checkpoint pathways.
* Major surgery within 28 days before the first experimental treatment (biopsy required for diagnosis is permitted).
* Subject with central nervous system (CNS) metastases.
* Had other active malignant tumors within 5 years before entering the study. Except for basal cell or squamous cell carcinomas, superficial bladder carcinomas, carcinoma in situ of the cervix, ductal carcinoma in situ, and papillary carcinoma of the thyroid, which may be treated locally and have been cured.
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis.
* The presence of clinically significant acute or chronic pancreatitis.
* The presence of other acute or chronic infections of clinically significant significance.
* History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
RP2D | Up to week 3
  Recommended Phase 2 Dose of SHR-1701
ORR | Up to approximately 6 months
  Objective Response Rate

SECONDARY OUTCOMES:
Clinically significant toxicity | Up to week 3
  above grade 3 AEs
OS rate | From the start of treatment to 9 months
  9-month-overall survival rate
AEs+SAEs | from the first drug administration to within 90 days for the last SHR-1701 dose
  Adverse Events and Serious Adverse Events
PFS | Up to approximately 6 months
  Progression-Free-Survival
DCR | Up to approximately 12 months
  Disease Control Rate
OS | up to 2 years
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai